CLINICAL TRIAL: NCT01189617
Title: A Single-center, Medically Supervised, Safety Evaluation Study of an All-in-One Body and Lubricant Product
Brief Title: Safety Study for an All-in-One Body and Personal Lubricant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Healthcare Products Division of McNEIL-PPC, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KOYNAP0011
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Lubricating Agents
Keywords: Personal Lubricant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Formula PD-F-7619 (Experimental): At least twice per week for one week, massage about a dime-sized amount of the PD-F-7619 personal lubricant product to the application site as directed.
  Interventions: Device: Formula PD-F-7619

INTERVENTIONS:
Device: Formula PD-F-7619 — Off-White to Beige Lotion
  Other Names: All-In-One Caressing Crème & Personal Lubricant; K-Y Touch Massage Warming 2-in-1 Personal Lubricant

SUMMARY:
This is a one-week study designed to test the safety of an all-in-one body and personal lubricant product during in-home use.

DETAILED DESCRIPTION:
This is a single-center, medically supervised, single-arm study to evaluate the safety of an all over body and personal lubricant product in home-use conditions via clinical assessment. The study will consist of 2 visits. Subjects who meet the entrance criteria will receive investigational product (IP) and 2 subjective questionnaires for at-home completion. The subjects will be required to use the IP at least 2 times, as instructed over the 1-week home-use period. At the end of the study (visit 2) subjects will return to the study site, at which time the unused IP and questionnaires will be returned and a final clinical assessment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy adults in a stable, monogamous, ongoing heterosexual relationship with current partner within protocol-specified parameters
* Subjects comfortable discussing sensitive topics such as personal hygiene, menstruation and sexuality
* Able to read and understand English
* Voluntarily signs an Informed Consent document after the trial has been explained
* Willing to follow all study procedures, including birth control requirements

Exclusion Criteria:

* Any medical or mental health history or condition, or use of any product, drug or medication that per protocol (or in the opinion of the Investigator) might compromise the participant's safety or the analysis of results
* Participation as a research subject in a different trial within timelines dictated by protocol
* Participants with relationships or employment outside protocol-defined parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherryl Frisch, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide; Melissa Israel, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- Concentrics Research, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Male: Male Participants
- Female: Female Participants
Period: Overall Study
Arm/Group | Male | Female
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (12.8) | 49.3 (12.8) | 50.25 (12.8)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 35 | 35
  Male | 35 | 0 | 35
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 21 | 25 | 46
  Black or African-American | 13 | 9 | 22
  American Indian or Alaska Native | 1 | 0 | 1
  Other [unknown] | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Female Sub-Typing - Menopausal State [Number; unit: Participants]
  Premenopausal | NA — Data for this element is not available for male subjects because they do not experience menopause. | 18 | 18
  Postmenopausal | NA — Data for this element is not available for male subjects because they do not experience menopause. | 17 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Irritation Score of "0" at Baseline and One Week
Description: Severity of irritation on a scale from 0 (No Irritation) to 6 (Presence of Lesions). Since a score of 0 is required at baseline for inclusion in the trial, this score represents a change from baseline and the trial is considered baseline-controlled.
Time Frame: Baseline and One Week
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 35 | 35
Participants
  Visit 1 - Baseline | 35 | 35
  Visit 2 - One Week | 35 | 35

ADVERSE EVENTS:
Time Frame: 1 Week (+30 days for Serious Adverse Events, and beyond if assessed as possibly treatment related)
Description: Subjects reported adverse events on questionnaires, and site staff recorded changes in medical status/history since study start. Itching, burning and stinging counted as adverse events.
Arm/Group | Male | Female
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Male (N=35) | Female (N=35)
Application Site Pain (burning, stinging) (General disorders) | 1 | 2
Application Site Erythema (redness) (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study is considered a work made for hire and the Sponsor retains all rights to publish results.